CLINICAL TRIAL: NCT05406089
Title: Effects of Short-term and Perioperative Antiviral Therapy on Prognosis After Hepatectomy for Hepatitis B Virus-related Hepatocellular Carcinoma
Brief Title: Effects of Antiviral Therapy on Patients With HBV-related HCC
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Hu Liangshuo, Principal Investigator, First Affiliated Hospital Xi'an Jiaotong University
Other Study IDs: No.XJTU1AF2021LSK-414
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-06

CONDITIONS: Hepatocellular Carcinoma; Hepatitis B Virus; Survival
Keywords: Hepatitis B virus; Antiviral therapy; Hepatectomy
MeSH Terms: conditions — Carcinoma, Hepatocellular; Hepatitis B | interventions — Pharmaceutical Preparations

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The short-term antiviral therapy (STAT) group: The short-term antiviral therapy (STAT) group was defined as individuals who received HBV antiviral ( antiviral treatments consisted of adefovir (10 mg/day), entecavir (0.5 mg/day), and lamivudine (100 mg/day) )at least 24 weeks before hepatectomy (antiviral therapy still continued during perioperative period). Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and characteristics of this group were collected and recorded for subsequent analysis.
  Interventions: Other: Medication history
- The perioperative antiviral therapy (PAT) group: The perioperative antiviral therapy (PAT) group was defined as individuals who received antiviral treatment perioperatively ( antiviral treatments consisted of adefovir (10 mg/day), entecavir (0.5 mg/day), and lamivudine (100 mg/day) ). Subjects matching the characteristics of this group were screened from the database according to inclusion and exclusion criteria, and characteristics of this group were collected and recorded for subsequent analysis.
  Interventions: Other: Medication history

INTERVENTIONS:
Other: Medication history — The study was retrospective and did not involve the application of interventions

SUMMARY:
Based on the follow-up data of patients who underwent hepatectomy for HBV-related HCC at the First Affiliated Hospital of Xi'an Jiaotong University. patients who met the enrollment criteria were screened for tumor recurrence and survival for statistical analysis to understand the prognosis of patients and analyze the risk factors affecting their prognosis.

DETAILED DESCRIPTION:
A retrospective study of patients who underwent hepatectomy for HBV-related HCC at the First Affiliated Hospital of Xi'an Jiaotong University from January 2016 to June 2019 was conducted. The clinical data of patients, including demographic features, perioperative laboratory values, surgical information, and pathological data, were collected from the official database for patients' data gathering, also, Based on the follow-up data of patients who met the enrollment criteria were screened for tumor recurrence and survival for statistical analysis to understand the prognosis of patients and analyze the risk factors affecting their prognosis.

ELIGIBILITY:
Inclusion Criteria:

Age of 18-70 years; Initial hepatectomy was performed; Positive HBsAg results and negative results for antibodies to hepatitis C virus (HCVAb) and human immunodeficiency virus; The patient did not undergo antitumor treatment, such as transcatheter arterial chemoembolization, radiofrequency ablation-chemotherapy or radiotherapy, or postoperative liver transplantation; Barcelona Clinic Hepatocellular carcinoma stage 0, A, or B (a few patients with stage C were also enrolled); Negative hepatectomy margin; No other tumors.

Exclusion Criteria:

Undergo antitumor treatment, such as transcatheter arterial chemoembolization, radiofrequency ablation-chemotherapy or radiotherapy, or postoperative liver transplantation; Positive results for antibodies to hepatitis C virus (HCVAb) and human immunodeficiency virus

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age 18 or older) who underwent hepatectomy between January 1st, 2016, and June 30st, 2019, were retrospectively identified using the database for clinical data in the First Affiliated Hospital of Xi'an Jiaotong University
Sampling Method: Non-Probability Sample
Enrollment: 494 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Post-operative survival time | Time from the end of hepatectomy to the patient's death, or the end of follow-up by December 31, 2020. whichever came first, assessed up to 60 months
  Postoperative survival time for patients receiving hepatectomy
Recurrence of the hepatocellular carcinoma after hepatectomy | The time period between hepatectomy and the initial examination revealing a recurrence of hepatocellular carcinoma, or until the end of follow-up on December 31, 2020.whichever came first, assessed up to 60 months.
  Recurrence of the hepatocellular carcinoma in patients who underwent hepatectomy

SECONDARY OUTCOMES:
Surgery information | Intraoperative
  Detailed information such as operation time

CONTACTS AND LOCATIONS:
Overall Officials: Bo Wang, MD PhD, Study Chair — First Affiliated Hospital Xi'an Jiaotong University

IPD SHARING:
Plan to Share IPD: No
The study was based on database from the The First Affiliated Hospital of Xi'an Jiao Tong University , researchers did not have access to patients' information nor raw data unless approved by the Ethics Committee of The First Affiliated Hospital of Xi'an Jiao Tong University.